CLINICAL TRIAL: NCT00451412
Title: A Randomized, Double-blind, Multi-center Comparison of the Efficacy and Safety of Certoparin (3000 U Anti-Xa o.d.) With Unfractionated Heparin (5000 IU t.i.d.) in the Prophylaxis of Thromboembolic Events in Acutely Ill Medical Patients
Brief Title: A Comparison of Certoparin and Unfractionated Heparin in the Prevention of Thromboembolic Events in Acutely Ill Medical Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CMEX839BDE03
Record Dates: First submitted 2007-03-21; First posted 2007-03-23 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-07

CONDITIONS: Thromboembolism
Keywords: Venous thromboembolism; Medical patients; Heparin; Low molecular weight heparin; Deep vein thrombosis; Certoparin; Embolism and Thrombosis
MeSH Terms: conditions — Thromboembolism; Venous Thromboembolism; Venous Thrombosis; Embolism and Thrombosis | interventions — certoparin; Sandoparin; heparin-dihydergot; Heparin, Low-Molecular-Weight; Heparin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Certoparin (Experimental)
  Interventions: Drug: Certoparin
- Unfractionated Heparin (Active Comparator)
  Interventions: Drug: Unfractionated Heparin

INTERVENTIONS:
Drug: Certoparin — 3000 U anti XA of certoparin in 0.3 ml solution, once daily
  Other Names: Sandoparin; Embolex; low molecular weight heparin
  Arms: Certoparin
Drug: Unfractionated Heparin — solution, 5000 IU of unfractionated heparin in 0.3 ml, 3 times daily
  Arms: Unfractionated Heparin

SUMMARY:
This study is designed to provide efficacy and safety data for certoparin in the prophylaxis of venous thromboembolism in immobilized, acutely ill medical patients.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized medical patients 70 years of age or older
2. Acute medical illness with significant decrease in mobility expected for at least 4 days (patient bedridden or only able to walk short distances)
3. written informed consent

Exclusion Criteria:

1. immobilization longer than 3 days prior to randomization
2. prior major surgery, trauma or invasive procedure within the last 4 weeks including any injuries or operation of central nervous system
3. expected major surgical or invasive procedure within the next 3 weeks after randomization
4. LMWH/heparin administration longer than 48 hours in the 5 days prior to randomization
5. immobilization due to cast or fracture
6. indication for anticoagulatory or thrombolytic therapy
7. acute symptomatic DVT / PE
8. known hypersensitivity to any of the study drugs or drugs with similar chemical structures
9. Acute or history of heparin induced thrombocytopenia type II (HIT II)

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 3254 (Actual)
Dates: Start 2007-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Incidence of venous thromboembolism during treatment (proximal deep vein thrombosis, pulmonary embolism, death related to venous thromboembolism) | 20 days

SECONDARY OUTCOMES:
proximal and distal deep vein thrombosis (DVT) (combined and separate) assessed by ultrasound screening, | 20 days
symptomatic DVT, | 20 days
symptomatic non-fatal pulmonary embolism (PE), | 20 days
combination of proximal DVT, non fatal PE and death from all causes including PE | 20 days
VTE related death, | 20 days

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- Novartis investigative sites, Nuremberg, Germany

REFERENCES:
- [Derived] Haas S, Schellong SM, Tebbe U, Gerlach HE, Bauersachs R, Melzer N, Abletshauser C, Sieder C, Bramlage P, Riess H. Heparin based prophylaxis to prevent venous thromboembolic events and death in patients with cancer - a subgroup analysis of CERTIFY. BMC Cancer. 2011 Jul 26;11:316. doi: 10.1186/1471-2407-11-316. PMID 21791091
- [Derived] Bauersachs R, Schellong SM, Haas S, Tebbe U, Gerlach HE, Abletshauser C, Sieder C, Melzer N, Bramlage P, Riess H. CERTIFY: prophylaxis of venous thromboembolism in patients with severe renal insufficiency. Thromb Haemost. 2011 Jun;105(6):981-8. doi: 10.1160/TH10-09-0614. Epub 2011 Apr 20. PMID 21505722
- [Derived] Tebbe U, Schellong SM, Haas S, Gerlach HE, Abletshauser C, Sieder C, Bramlage P, Riess H. Certoparin versus unfractionated heparin to prevent venous thromboembolic events in patients hospitalized because of heart failure: a subgroup analysis of the randomized, controlled CERTIFY study. Am Heart J. 2011 Feb;161(2):322-8. doi: 10.1016/j.ahj.2010.10.005. PMID 21315215